CLINICAL TRIAL: NCT03446742
Title: Effectiveness of Stratification Protocols and Clinical, Physical and Biochemical Parameters to Forecast Intercurrences in Cardiovascular Rehabilitation Programs.
Brief Title: Stratification Protocols and Clinical, Physical and Biochemical Parameters to Forecast Cardiovascular Intercurrences.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Other Study IDs: 79213417.0.0000.5402
Record Dates: First submitted 2018-01-29; First posted 2018-02-27 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Rehabilitation Service; Signals and symptons; Heart Rate; Blood pressure; Respiratory Muscles; autonomic modulation; exercise; risk measurement; muscle strength; inflammation; cytosines
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Inflammation | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiovascular rehabilitation group: Initially all patients will have their charts analyzed, from which data will be extracted for characterization of the population, and anthropometric data will be measured for calculation of body mass index. Afterwards, patients will have their clinical, physical and biochemical parameters. They will be followed up for a period of 2 months during the routines of the cardiovascular rehabilitation sessions for assessment of signs and symptoms. In the second stage the patients will perform the normal routines of their cardiovascular rehabilitation program for a period of 6 months. In the third stage, patients will have their clinical, physical and biochemical parameters and then followed up for another 2 months during the routines of the sessions of the cardiovascular rehabilitation program to evaluate signs and symptoms, which will allow to evaluate if gains/losses in the physical parameters can exert influences in the appearance of signs and symptoms during the sessions.
  Interventions: Other: Cardiovascular rehabilitation

INTERVENTIONS:
Other: Cardiovascular rehabilitation — The cardiovascular rehabilitation program is performed three times weekly on alternate days and each session lasts approximately 60 minutes divided as follows: 5 minutes to the initial rest where blood pressure (BP), heart rate (HR) and signs and symptoms are assessed; 15 minutes of warm-up, composed by global stretches, lower and upper limb exercises, and exercises combining the two modes; then, patients go to the resistance phase (30 minutes), where are performed an individualized aerobic protocol according to their HR reserve values using bicycle and treadmill (at the 4th and 10th minute of both ergometers at HR is evaluated, and in the bicycle is also evaluated the BP of all the patients). The end of the protocol is composed of 10-minute relaxation, during which the patients perform a small cardiovascular deceleration (a few laps around the room, with free speed) and, finally, lie down at rest. The presence of signs and symptoms is assessed at all stages of the program.

SUMMARY:
Introduction: Despite the various beneficial effects, cardiovascular rehabilitation programs (CVRP) have been associated with the appearance of signs and symptoms. Risk stratification protocols are used to stratify into risk trials for an occurrence of events during physical exercise, although studies investigating their efficacy in predicting signs and symptoms during VCTV are inconclusive. In addition, several clinical, physical and biochemical parameters have been used in the literature as risk markers for the appearance of adverse events, and to investigate whether these parameters are capable of predicting a possibility of intercurrences during PRCV sessions.Objectives: 1) to evaluate the efficacy of risk stratification protocols in predicting signs and symptoms during the performance of a PRCV; 2) to analyze the correlation between clinical, physical and biochemical parameters measured at rest with the presence of signs / symptoms in participants of a PRCV; 3) to evaluate whether changes in clinical, physical or biochemical parameters induced by PRCV influence the appearance of signs and symptoms during PRCV. Materials and Methods: To perform this study, data from 70 patients inserted in a PRCV will be evaluated. The study will be divided into three subprojects that can be divided into three stages: 1) risk stratification of patients who will participate in the study by two independent evaluators (Study 1) and evaluation of clinical parameters (cardiorespiratory parameters and autonomic modulation evaluation); (maximal isometric resistance, maximal isometric contraction, functional capacity and level of physical activity) and biochemical (IL-6, TNF-alpha and IL-10) (Studies 2 and 3). Patients will then be followed up by 24 sessions during the PRCV routines to evaluate signs and symptoms, for posterior correlation with the risk stratification obtained in each protocol (Study 1), and with resting values of clinical, physical and biochemical studies (Studies 2 and 3); 2) Patients perform the normal routines of their PRCV for a period of 6 months (Study 3); 3) The patients will again have their clinical, physical and biochemical parameters evaluated and then will be followed up for another 2 months (24 sessions) during the routines of the PRCV sessions to evaluate signs and symptoms, which will allow to evaluate if gains / losses in these parameters exert influence on the appearance of signs and symptoms during PRCV sessions.

ELIGIBILITY:
Inclusion Criteria:

* To present clinical diagnosis of cardiovascular disease and/or cardiovascular risk factors;
* Be able to perform all the proposed evaluations;
* Agree to participate in the studies.

Exclusion Criteria:

* Patients who miss more than six consecutive sessions of the program or those who total more than 12 absences during the two months that total the period of analysis of the signs and symptoms will be excluded from the analyzes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals, regardless of gender, who participate in the cardiovascular rehabilitation program developed at the Center for Studies and Attendance in Physiotherapy and Rehabilitation of the São Paulo State University.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Autonomic modulation | 6 months
  The autonomic modulation will be evaluated by heart rate variability method
Blood pressure | 6 months
  The blood pressure will be evaluated with a non invasive method
Heart rate | 6 months
  The heart rate will be evaluated with an pulse oximeter with the volunteers at rest
Spirometric parameters | 6 months
  The spirometric parameters will be evaluated by spirometry method.
Maximum expiratory and inspiratory pressure | 6 months
  The maximum expiratory and inspiratory pressure will be evaluated by manovacuometry method.
maximum isometric muncle strength | 6 months
  The vollunteers will realize the maximum isometric strength with a dominant member during 5 seconds, and the maximum value obtained will be registered.
voluntary isometric contraction | 6 months
  The volunteers will do a maximum voluntary isometric contraction and instructed to maintain this contraction as longer they can. The maximum time obtained will be registered.
Cardiorrespiratory fitness | 6 months
  The vollunters will be submited to a maximum effort test to define their cardiorrespiratory fitness.
Physical activity level | 6 months.
  The physical activity of the volunteers will be registered during one week to determine their physical activity level.
Biochemical parameters | 6 months
  Inflamatory (TNF-alpha, IL-6) and anti-inflamatory cytokines (IL-10) will be analysed by blood samples.
Cardiovascular risk stratification protocols | 2 months
  The cardiovascular risk stratification will be evaluated by seven diferent protocols and the volunteers will be stratified like less, medium and high cardiovascular risk. There will be used protocols of the organizations below: American College of Sports Medicine, Sociedade Brasileira de Cardiologia, American Heart Association, Frederic J. Pashkow protocol, American Association of Cardiovascular and Pulmonary Rehabilitation, Société Française de Cardiologie and Sociedad Española de Cardiología
Cardiovascular signals | 6 months
  Signals like pulse rate changes, increased SBP and DBP during exercise, tachipnea, pallor will be observed by the evaluator and the presence or absence will be registered.
Cardiovascular symptoms | 6 months
  Symptoms like dizziness, angina pectoris, cramp, muscle pain, fatigue, nausea will be related for the volunteers, and the presence or absence will be registered.

SECONDARY OUTCOMES:
oxygen saturation | 6 months
  The respiratory parameter oxigen saturation of the volunteers will be evaluated with a pulse oximeter with the volunteers at rest.
Respiratory frequency | 6 months
  The respiratory parameters respiratory frequency will the evaluated by number of tract per minute with the volunteers at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos M Vanderlei, PhD, Study Director — Universidade Estadual Paulista - UNESP campus de Presidente Prudente

IPD SHARING:
Plan to Share IPD: No
I don't have plans.

REFERENCES:
- [Derived] Ribeiro F, Takahashi C, Vanzella LM, Laurino MJL, Lima IM, Silva VEDS, Silva JPLN, Valente HB, da Silva AKF, Christofaro DGD, Vanderlei LCM. An investigation into whether cardiac risk stratification protocols actually predict complications in cardiac rehabilitation programs? Clin Rehabil. 2021 May;35(5):775-784. doi: 10.1177/0269215520978499. Epub 2020 Dec 8. PMID 33292000
- [Derived] Vanzella LM, Takahashi C, Ribeiro F, Lima IM, Silva AKFD, Christofaro DGD, Vanderlei LCM. Efficacy of risk stratification protocols and clinical, physical, and biochemical parameters to previse signals and symptoms during cardiovascular rehabilitation programs: Protocol for an observational trial. Medicine (Baltimore). 2019 Jun;98(24):e15700. doi: 10.1097/MD.0000000000015700. PMID 31192910